CLINICAL TRIAL: NCT06011720
Title: Collaborative Study to Reduce Length of Stay and Improve Transitions of Care for Stroke Patients at Robert Wood Johnson University Hospital & JFK Johnson Rehabilitation Institute
Brief Title: Transitions of Care for Stroke Patients
Status: Recruiting | Type: Observational
Sponsor: Kiwon Lee MD (Other)
Collaborators: JFK Medical Center (Other)
Responsible Party: Sponsor-Investigator, Kiwon Lee MD, Professor of Neurology, Rutgers, The State University of New Jersey
Organization: Rutgers, The State University of New Jersey (Other)
Other Study IDs: Pro2019000095
Record Dates: First submitted 2022-02-18; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Stroke; Ischemic Stroke; Intracerebral Hemorrhage
Keywords: Stroke; physiatry; rehabilitation; PM&R consultation; Transient Ischemic Attack; Intracerebral Hemorrhage; Ischemic Stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke; Cerebral Hemorrhage; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke Patients July 1st 2015 - June 30th 2017: Stroke patients that have undergone hospitalization within the time frame July 1st 2015 - June 30th 2017 to be used as a baseline.
- Stroke Patients January 1st 2018 - December 31st 2019: Stroke patients that have undergone hospitalization and undergone improvements to transition of care within the time frame January 1st 2018 - December 31st 2019.
  Interventions: Other: Improved transition of care.

INTERVENTIONS:
Other: Improved transition of care. — Evaluation of how early physiatry consultation after acute stroke affects length of stay and resulting outcomes.
  Groups: Stroke Patients January 1st 2018 - December 31st 2019

SUMMARY:
For stroke patients, early initiation of therapy typically yields the best functional outcomes. Rehabilitation of stroke patients immediately after hospitalization minimizes deleterious effects of immobility and facilitates restoration of function. The investigators are testing if coordinated efforts between the medical and rehabilitation disciplines may improve stroke patient's functional recovery and subsequent follow-ups after discharge.

DETAILED DESCRIPTION:
Stroke is the fifth leading cause of mortality, claiming the lives of 133,000 individuals in the United States annually. Approximately one-quarter of the 795,000 annual strokes are recurrent. It is estimated that up to 80% of all strokes can be prevented. Forty percent of stroke survivors sustain moderate functional impairments and 15% to 30% sustain severe disability. Approximately 25% of adult stroke patients are readmitted to the hospital within six to twelve months of their preliminary stroke. Identifying and implementing effective medical and rehabilitation interventions is critical in providing care to stroke patients. The goal is to provide optimal, cost-effective care that: 1) prevents secondary medical complications, readmissions, and recurrent disease, and 2) maximizes patient function physically, cognitively, and socially. JFK Johnson Rehabilitation Institute (JRI) proposes a collaborative study with Robert Wood Johnson University Hospital (RWJUH) that addresses this issue while proving beneficial to stroke patients at both institutions. Streamlining the physiatry consult process will improve access to rehabilitation medicine specialty care for acute patients at RWJUH and help facilitate the transfer of stroke patients to the next most appropriate level of care.

ELIGIBILITY:
Inclusion Criteria:

* Stroke patients hospitalized within Robert Wood Johnson University Hospital system for Ischemic Stroke or Intracerebral Hemorrhage.

Exclusion Criteria:

* Those not in the Robert Wood Johnson University Hospital system.
* Those with a Subarachnoid Hemorrhage or Transient Ischemic Attack (< 24 hours).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients hospitalized within Robert Wood Johnson University Hospital system for Ischemic Stroke or Intracerebral Hemorrhage within the two time frames, July 1st 2015 - June 30th 2017 and January 1st 2018 - December 31st 2019.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Length of stay (in hours and days). | Data from 1/1/2018-12/31/2019, collected under updated standard of care compared to baseline data from 7/1/2015-6/30/2017.
  We standardized the placement of early physiatry consults during patient admission. We will determine the effect this has on overall acute care length of stay in ischemic and hemorrhagic stroke patients.

SECONDARY OUTCOMES:
Rehospitalization rate. | Data from 1/1/2018-12/31/2019, collected under updated standard of care compared to baseline data from 7/1/2015-6/30/2017.
  We standardized placement of early physiatry consults during patient admission, and will determine the effect this has on acute care readmission rates (for the same stroke related problems). This will be measured as absolute value and mean number of readmissions in the preintervention group and the post-intervention group, as well as percent of patients with readmissions in each group.
Functional independence | Data from 1/1/2018-12/31/2019, collected under updated standard of care compared to baseline data from 7/1/2015-6/30/2017.
  We standardized placement of early physiatry consults during patient admission, and will determine any differences in long term functional independence by means of a 90 day modified Rankin Scale (mRS) - a standard rater driven scale that characterizes patient's level of independence on a scale of 0-6 (0 being without symptoms and 6 being deceased).
Stroke clinic outpatient follow-up. | Data from 1/1/2018-12/31/2019, collected under updated standard of care compared to baseline data from 7/1/2015-6/30/2017.
  We standardized placement of early physiatry consulted during patient admission, and will determine the rate of stroke clinic outpatient follow-up, as measured by absolute number of patients who follow-up at least once. We will further determine the relative percentage of patients who follow-up in stroke clinic for the preintervention and postintervention group.
Pre-specified subanalyses for effect on primary outcome measures. | Data from 1/1/2018-12/31/2019, collected under updated standard of care compared to baseline data from 7/1/2015-6/30/2017.
  We will assess the independent effects of multiple variables on length of stay, functional independence and stroke clinic outpatient follow-up. The pre-specified variables include: presence/number/nature of medical comorbidities, stroke type (i.e. ischemic vs. hemorrhagic), insurance type (i.e. private insurance, Medicaid, managed Medicaid, etc.), severity of stroke on admission (measured by NIHSS or ICH score), prior antithrombotic use.
Pre-specified subanalyses for effect on functional independence. | Data from 1/1/2018-12/31/2019, collected under updated standard of care compared to baseline data from 7/1/2015-6/30/2017.
  We will assess the independent effects of multiple variables on functional independence (mRS). The variables include: time between discharge and rehab admittance (days and hours), rehab length of stay (days and hours), and presence of outpatient follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Kiwon Lee, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Rutgers-RWJMS Department of Neurology, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No